CLINICAL TRIAL: NCT00618774
Title: An Open-label, Long-term Study of Telmisartan Plus Amlodipine Fixed-dose Combination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1235.16
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Drug: telmisartan40/amlodipine5
Drug: telmisartan80/amlodipine5

SUMMARY:
To assess the long term safety and efficacy of telmisartan plus amlodipine FDC in patients with essential hypertension who failed to control their BP with either monotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension
2. Outpatient

Exclusion Criteria:

* Patients whose SBP >=180 mmHg or DBP >=110 mmHg at the end of treatment visit of the double-blind treatment period in the "non-responder trials"
* Patients who have met any of the exclusion criteria defined in the "non-responder trials"

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Japan (7):
  - 1235.16.004 Boehringer Ingelheim Investigational Site, Chofu, Tokyo
  - 1235.16.006 Boehringer Ingelheim Investigational Site, Nishi-ku, Hiroshima, Hiroshima
  - 1235.16.005 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1235.16.007 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1235.16.003 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1235.16.001 Boehringer Ingelheim Investigational Site, Shinjyuku-ku,Tokyo
  - 1235.16.002 Boehringer Ingelheim Investigational Site, Suita, Osaka

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Started | 211 | 48
Completed | 205 | 45
Not Completed | 6 | 3
Not completed — Adverse Event | 5 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination | Total
Number analyzed (Participants) | 211 | 48 | 259
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.8 (9) | 51.1 (8) | 55.8 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 4 | 54
  Male | 161 | 44 | 205

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Adverse Events
Description: An adverse event is defined as any untoward medical occurrence
Time Frame: 52 weeks
Population: Treated set for safety, which was the analysis set including all the patients who had valid measurements after drug administration.
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 211 | 48
percentage of participants | 77.3 | 77.1

2. Secondary Outcome: Change From Baseline in Seated Diastolic Blood Pressure at Week 8
Description: mean reduction from pseud-baseline (after the washout) in seated diastolic blood pressure
Time Frame: Baseline and week 8
Population: Full analysis set for blood pressure measurements, which was the analysis set including all the patients who had valid measurements at the reference baseline and at one or more time-points after reference baseline.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
mmHg | 20.81 (6.65) | 15.75 (6.61)

3. Secondary Outcome: Change From Baseline in Seated Systolic Blood Pressure at Week 8
Description: mean reduction from pseud-baseline (after the washout) in seated systolic blood pressure
Time Frame: Baseline and week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
mmHg | 33.89 (12.2) | 26.44 (11.68)

4. Secondary Outcome: Seated DBP Control Rate at Trough After 8 Weeks
Description: Percentage of patients whose DBP <90 mmHg after 8 weeks of treatment
Time Frame: week 8
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
percentage of participants | 91.8 | 52.1

5. Secondary Outcome: Seated SBP Control Rate at Trough After 8 Weeks
Description: Percentage of patients whose SBP <140 mmHg after 8 weeks of treatment
Time Frame: Week 8
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
percentage of participants | 93.2 | 85.4

6. Secondary Outcome: Change From Baseline in Seated Diastolic Blood Pressure
Description: Mean reduction from pseud-baseline (after the washout) in seated diastolic blood pressure
Time Frame: Baseline and week 20 / week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
mmHg
  Week 20 | 20.67 (7.16) | 16.36 (5.93)
  Week 48 | 21.39 (6.6) | 17.78 (7.31)

7. Secondary Outcome: Change From Baseline in Seated Systolic Blood Pressure
Description: mean reduction from pseud-baseline (after the washout) in seated systolic blood pressure
Time Frame: Baseline and week 20 / week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
mmHg
  Week 20 | 33.73 (12.55) | 27.18 (11.83)
  Week 48 | 33.97 (11.75) | 28.11 (12.78)

8. Secondary Outcome: Seated DBP Control Rate at Trough After 6 and 12 Months
Description: Percentage of patients whose DBP <90 mmHg.
Time Frame: 6 months and 12 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
percentage of participants
  Week 20 | 90.8 | 54.2
  Week 48 | 92.8 | 66.7

9. Secondary Outcome: Seated SBP Control Rate at Trough After 6 and 12 Months
Description: Percentage of patients whose SBP <140 mmHg
Time Frame: 6 months and 12 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
percentage of participants
  Week 20 | 95.7 | 89.6
  Week 48 | 93.2 | 89.6

10. Secondary Outcome: Seated DBP Response Rate at Trough
Description: Percentage of patients whose DBP <90 mmHg or decreased from pseudo-baseline by >=10 mmHg at 6 months and 12 months
Time Frame: 6 months and 12 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
percentage of participants
  Week 20 | 97.1 | 85.4
  Week 48 | 98.6 | 87.5

11. Secondary Outcome: Seated SBP Response Rate at Trough
Description: Percentage of patients whose SBP <140 mmHg or decreased deom pseudo-baseline by >=20 mmHg after 6 and 12 months
Time Frame: 6 months and 12 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
percentage of participants
  Week 20 | 97.6 | 93.8
  Week 48 | 97.6 | 93.8

12. Secondary Outcome: Seated Blood Pressure Normalisation at Trough
Description: Percentage of patients when classifying their blood pressure measurements into the following classes at 6 and 12 months:
  Optimal: SBP <120 mmHg and DBP <80 mmHg
  Normal: SBP >=120 mmHg or DBP >=80 mmHg and SBP <130 mmHg or DBP <85 mmHg
  High normal: SBP >=130 mmHg or DBP >=85 mmHg and SBP <140 mmHg or DBP <90 mmHg
  No: SBP >=140 mmHg or DBP >=90 mmHg
Time Frame: 6 months and 12 months
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 207 | 48
percentage of participants
  Week 20: Optimal | 29.5 | 4.2
  Week 20: Normal | 35.3 | 18.8
  Week 20: High Normal | 24.2 | 31.3
  Week 20: No | 11.1 | 45.8
  Week 48: Optimal | 32.4 | 6.3
  Week 48: Normal | 36.2 | 18.8
  Week 48: High Normal | 18.4 | 39.6
  Week 48: No | 13.0 | 35.4

13. Primary Outcome: Clinically Relevant Abnormalities for Changes in Blood Pressure and Pulse Rate Due to Position Change, Seated Pulse Rate, Laboratory Parameters and ECG
Description: Clinically relevant abnormalities for changes in blood pressure and pulse rate due to position change, seated pulse rate, laboratory parameters and ECG. New abnormal findings or worsening of baseline conditions were reported as adverse events.
Time Frame: First administration of study treatment to 24 hours post last dosing of study treatment.
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Number analyzed (Participants) | 211 | 48
participants
  Blood Pressure Decreased | 2 | 0
  Prostatic specific antigen increased | 1 | 0
  Acute myocardial infarction | 0 | 1
  Arrhythmia | 1 | 0
  Atrial fibrillation | 2 | 0
  Extrasystoles | 1 | 0
  Ventricular extrasystoles | 1 | 0
  Orthostatic hypotension | 0 | 1

ADVERSE EVENTS:
Time Frame: While being treated with T20+A5, T40/A5, T80/A5, T40/A5+additional treatment, T80/A5+additional treatment and within 24 hours from the last dosing of any of them.
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination
Serious Adverse Events (participants affected / at risk) | 9/211 | 3/48
Other Adverse Events (participants affected / at risk) | 102/211 | 23/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination (N=211) | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination (N=48)
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination (N=211) | Telmisartan 80 mg Plus Amlodipine 5 mg Fixed-dose Combination (N=48)
Dental caries (Gastrointestinal disorders) | 12 | 3
Nasopharyngitis (Infections and infestations) | 91 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.